CLINICAL TRIAL: NCT06575712
Title: Coping Skills Training for Symptom Management and Daily Steps (Step Up)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00116334
Record Dates: First submitted 2024-08-15; First posted 2024-08-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Stem Cell Transplant; CAR-T Cell Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Up (Experimental): Step Up participants will complete 7 sessions over 7-14 weeks (45 min/session). Of the 7 sessions, participants will complete 3 in-person in the hospital/outpatient clinic (1 coping skills training for symptom management [45 min] and 2 activity coaching [45 min]) followed by 4 via videoconferencing (coping skills training for symptom management and activity coaching [45 min each]) once the patient has been discharged home from the outpatient clinic.
  Interventions: Behavioral: Step Up
- Usual Care Plus (UC+) (Other): Usual Care Plus (UC+) participants will complete all assessments at time intervals corresponding to Step Up, and otherwise continue to receive their usual medical care plus 7 videos delivering educational content (1 video/week for 7 weeks; 5-10 minutes/video) via a study app (free download), but not the Step Up protocol.
  Interventions: Other: Usual Care Plus (UC+)

INTERVENTIONS:
Behavioral: Step Up — A hybrid in-person and mHealth (mobile health) coping skills training and activity coaching intervention.
  Arms: Step Up
Other: Usual Care Plus (UC+) — Usual medical care plus videos delivering educational content via an app.
  Arms: Usual Care Plus (UC+)

SUMMARY:
The aim of this study is to test the efficacy of a hybrid in-person and mHealth coping skills training and activity coaching intervention (Step Up), to enable HCT patients to effectively cope with symptoms (pain, fatigue, and stress) to improve their ability to engage in physical activity that can improve physical disability.

DETAILED DESCRIPTION:
The objective of this R01 project is to use novel mobile health (mHealth) behavioral intervention approaches to enable patients who have undergone hematopoietic stem cell transplant (HCT) and Car T cell therapy to effectively cope with their symptoms to improve their ability to engage in physical activity that can improve physical disability. In a NCI R21 study, we developed a hybrid in-person and mHealth Coping Skills Training for Symptom Management and Daily Steps (Step Up) intervention protocol, including mobile app. Step Up provides HCT and CAR T patients with cognitive behavioral coping skills training and occupational therapy (OT)-led activity coaching sessions to enhance their ability to cope with symptoms - fatigue, pain, distress - that interfere with physical activity. Step Up has been developed by experts in symptom management, members of the HCT medical team, and with extensive input from HCT patients. Our R21 results show Step Up is feasible, acceptable to patients, and demonstrates a strong signal for intervention benefits, including improvements in physical disability, symptoms, and activity (daily steps). This R01 project uses a randomized controlled trial (RCT) to test the efficacy of Step Up compared to Usual Care Plus (UC+). Step Up includes a mobile app and activity trackers (Garmins) to capture daily symptom, activity, and biometric data allowing the study team to provide real-time personalized feedback. Our central hypothesis is Step Up will lead to improvements in physical disability (primary outcome), as well as secondary outcomes of symptom severity, physical activity, and digital biomarkers reflective of symptom burden following HCT. A RCT (N=177) will be used to pursue three specific aims: 1) Test the efficacy of Step Up for improving physical disability, as well as symptom severity, physical activity, and self-efficacy for symptom management compared to UC+; 2) Examine the relationship between symptoms and activity; and 3) Test the efficacy of Step Up for improving digital biomarkers reflective of symptom burden (heart rate, activity, sleep time) measured via Garmins. The proposed work is innovative and impactful for HCT and CAR T patients as it addresses interfering symptoms, integrates evidence-based coping skills training with OT sessions to increase activity while decreasing symptoms that interfere with activity, and uses mHealth technology for personalized real-time feedback to patients. Positive results would provide the first demonstration of efficacy of a hybrid-delivered cognitive behavioral coping skills training and activity coaching intervention that reduces physical disability by concurrently and synergistically decreasing symptom burden and increasing activity. The proposed research has the potential to produce significant public health benefit by redesigning existing modes of behavioral intervention delivery, improving continuity and coordination of care, and ultimately enhancing patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* receipt of an autologous (auto) HCT or CAR-T cell therapy due to a hematologic malignancy, such as a diagnosis of leukemia, lymphoma, multiple myeloma
* age >18
* self-reported fatigue, pain, and psychological distress (confirmed at recruitment) - minimum two of three symptoms reported at >3 on 0-10 scale
* life expectancy > 12 months

Exclusion Criteria:

* cognitive impairment (e.g., dementia) recorded in the chart or suspected by provider
* metastases to the brain
* presence of a severe psychiatric condition (e.g., psychotic disorder) that would contraindicate safe participation as indicated by the medical chart, treating oncologist, or interactions with the medical/study staff
* inability to converse in English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical disability as measured by the Functional Assessment of Cancer Therapy (FACT) | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  The FACT is widely used in oncology research and includes four subscales assessing physical, functional, social/family, and emotional well-being. The 7-item physical subscale will be used in this study to assess physical disability. Each item is rated on a 5-point Likert scale (0 to 4). The total score is the sum of all items and thus ranges from 0 to 28, where higher scores indicate better physical well-being.
Change in physical disability as measured by the Six-Minute Walk Test (6MWT) | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  A self-paced timed walk test, the 6MWT is sensitive to change following medical treatments and has shown moderate correlations with physical disability. It measures the distance a patient walks in 6 minutes.

SECONDARY OUTCOMES:
Change in fatigue as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Adult Fatigue Profile 6-item Short Form | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  Fatigue will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Adult Fatigue Profile 6-item Short Form. The PROMIS F-SF consists of seven items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 = never to 5 = always. One item, "How often did you have enough energy to exercise strenuously," is reverse scored. The total score is used in the analysis and is obtained by summing keyed scores of all items. Scores can range from 7 to 35, with higher scores indicating greater fatigue.
Change in pain as measured by the 4-item Brief Pain Inventory (BPI) | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  The BPI is a scale used to rate pain severity and interference over the last 7 days. Pain severity is rated on a scale from 0=no pain to 10=worst pain imaginable in response to "average pain", "worst pain", "least pain", and "pain right now". An average of the responses to these four items is used to create a single pain severity score where higher scores indicate greater pain. Pain interference is rated on a scale from 0=does not interfere to 10=completely interferes in response to how much pain has interfered with different areas of life.
Change in psychological distress as measured by the Brief Symptom Inventory (BSI) | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  The BSI-18 will be condensed to include 12 items. Responses are rated on a 5-point scale where 0=not at all and 4=extremely. The total score ranges from 0 to 48, where higher scores indicate greater distress.
Change in activity as measured by daily step count | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  Step count will be measured by a Garmin Vivosmart 5 activity tracker that has a 6+ day battery life, syncs wirelessly and automatically to computers and smartphones, and resets at midnight. Garmins automatically sync daily with the study app.
Change in self-efficacy for managing symptoms as measured by the PROMIS Self-Efficacy for Managing Symptoms 8-Item Short Form | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  The PROMIS Self-Efficacy for Managing Symptoms 8-Item Short Form inquires about participants' level of confidence in their ability to manage symptoms. Responses are on a 5-point Likert scale where 1=I am not at all confident to 5=I am very confident. The total summed score ranges from 8 to 40, where higher scores reflect more self-efficacy.
Pre-Existing Physical Activity Behavior will be measured using the Stanford Leisure-Time Activity Categorical Item (L-Cat) | Baseline, Post-Intervention (2-3 months after Baseline), 3-month Follow-Up, 6-Month Follow-Up
  Participants identify which category best describes their level of activity during leisure time in the last month. Categories range from 0 "inactive" to 5 "very active."

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No